CLINICAL TRIAL: NCT04221854
Title: Stool-based SDC2 DNA Methylation Test vs. Fecal Immunochemical Test on the Detection of Colorectal Advanced Adenomatous Polyps and Cancer in Chinese Population: A Multi-central Randomized Clinical Trial
Brief Title: Stool-based SDC2 DNA Methylation Test for the Detection of Colorectal Advanced Adenomatous Polyps and Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Shanghai Municipal Center for Disease Control and Prevention (Other); Changhai Hospital (Other); Tianjin Nankai Hospital (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Guangzhou Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Ping Lan, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CCRCSIP
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer; Colorectal Adenomatous Polyp; Screening
Keywords: Colorectal cancer screening; SDC2 DNA Methylation; Fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will received either Stool-based SDC2 DNA Methylation Test or Fecal Immunochemical Test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stool-based SDC2 DNA methylation test group (Experimental): Subjects will received the stool-based SDC2 DNA methylation test for the screening of colorectal advanced adenomatous polyps and cancer.
  Interventions: Diagnostic Test: Stool-based SDC2 DNA methylation test
- Fecal immunochemical test group (Active Comparator): Subjects will received the fecal immunochemical test for the screening of colorectal advanced adenomatous polyps and cancer.
  Interventions: Diagnostic Test: Fecal immunochemical test

INTERVENTIONS:
Diagnostic Test: Stool-based SDC2 DNA methylation test — Stool-based SDC2 DNA methylation test
  Arms: Stool-based SDC2 DNA methylation test group
Diagnostic Test: Fecal immunochemical test — Fecal immunochemical test
  Arms: Fecal immunochemical test group

SUMMARY:
The primary objective is to compare the performance of Stool-based SDC2 DNA Methylation Test and commercially available Fecal Immunochemical Test(FIT) , on the detection rate of advanced adenomatous polyps and colorectal cancer in Chinese population. Subjects with positive results in either test will receive colonoscopy. Lesions will be confirmed as malignant or precancerous by colonoscopy and histopathologic examination.

DETAILED DESCRIPTION:
A large cohort of participants will be asked to collect stool sample for either Stool-based SDC2 DNA Methylation Test or Fecal Immunochemical Test. Subjects who have positive results will undergo colonoscopy within 6 months.

Representative histopathology slides from tissue biopsied or excised during colonoscopy and those from subsequent definitive surgery may be retrieved in order to be evaluated by pathologists to confirm the diagnosis and staging.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is average risk for development of colorectal cancer.
2. Subject is able and willing to undergo a screening colonoscopy within six months of enrollment.
3. Subject is 45 to 80 years of age inclusive.
4. Subject is able to comprehend, sign, and date the written informed consent document to participate in the study.
5. Subject is able and willing to provide stool samples according to written instructions provided to them.

Exclusion Criteria:

1. Subject has any condition which, in the opinion of the investigator should preclude participation in the study.
2. Subject has a history of colorectal cancer or adenoma.
3. Subject has a history of other digestive tract cancer.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The Detection Rate of Colorectal Polyps, Advanced Adenomatous Polyps and Cancer by Two Screening Methods | One year
  The stool-based SDC2 DNA methylation test CT values of 38 or less compared to beta-actin considered to be positive. Fecal immunochemical test values of more than 100 ng of hemoglobin per milliliter of buffer were considered as positive. An optical colonoscopy is used as diagnostic method. Lesions will be confirmed by histopathologic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Gu, MD, Principal Investigator — Shanghai Municipal Center for Disease Control and Prevention; Enda Yu, MBBS, Principal Investigator — Changhai Hospital; Ximo Wang, MD, PhD, Principal Investigator — Tianjin Nankai Hospital; Shan Wang, MD, PhD, Principal Investigator — Peking University People's Hospital; Jiahua Leng, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; Dong Xu, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Pengzhe Qin, MD, Principal Investigator — Guangzhou Center for Disease Control and Prevention
Locations (8):
- China (8):
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Beijing Cancer Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Guangzhou Center for Disease Control and Prevention, Guangzhou
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Changhai Hospital, Shanghai
  - Shanghai Municipal Center for Disease Control and Prevention, Shanghai
  - Tianjin Nankai Hospital, Tianjin

REFERENCES:
- [Derived] Chen Y, Li J, Gu K, Ding K, Qin P, Pei Z, Gong Y, Xu D, Liang Y, Yang D, Dou J, Huang Y, Hu J, Wu P, Zhang S, Wang W, Shi L, Liu Q, Li C, Li W, Wang X, Lan P, Liang B, He X. Stool-based methylated syndecan-2 test and fecal immunochemical test for advanced colorectal neoplasia screening in the Chinese population: A multicenter randomized noncomparative study. Chin Med J (Engl). 2025 Dec 3. doi: 10.1097/CM9.0000000000003897. Online ahead of print. PMID 41334638